CLINICAL TRIAL: NCT06251102
Title: Real-world Ruxolitinib Experience in Polycythemia Vera: REVIEW Study
Brief Title: Real-world Ruxolitinib Experience in PV
Acronym: REVIEW
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: MPN0224
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Polycythemia Vera
Keywords: ruxolitinib
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentric, observational, retro-prospective study in adult PV patients - resistant or intolerant to hydroxyurea - who are going to receive or have already initiated treatment with ruxolitinib according to the approved local label. Enrolment will last 9 months after the first enrolled patient. Patients will be observed for a minimum of 3 months, in order to evaluate the primary endpoint for all patients.

DETAILED DESCRIPTION:
This is a multicentric, observational, retro-prospective study in adult population who have been diagnosed with polycythemia vera according to the 2022 (WHO or ICC) criteria, who are resistant or intolerant to hydroxyurea and who are going to be prescribed or have already initiated treatment with ruxolitinib according to the approved local label. Patients who started treatment with ruxolitinib - according to clinical practice - will be enrolled. Enrolment will last 9 months after the first enrolled patient. Patients will be observed for a minimum of 3 months, in order to evaluate the primary endpoint for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years of age
2. Subjects must be diagnosed with PV according to the 2022 World Health Organization (WHO) or International Consensus Classification (ICC) criteria
3. Subjects must have a treatment history for PV that meets the definition of resistance or intolerance to hydroxyurea (HU) in accordance with the indications of the Italian Medicines Agency
4. Patients already on ruxolitinib treatment (retrospective cohort) at the start date of the study or patients who will start ruxolitinib (prospective cohort) during the study enrollment
5. Signed informed consent

Exclusion Criteria:

1. Different diagnosis from PV [eg. other chronic myeloproliferative neoplasia such as essential thrombocythemia, myelofibrosis; or of congenital erythrocytosis or secondary erythrocytosis]

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Polycythemia vera according to WHO or ICC 2022 criteria who received treatment with ruxolitinib as second-line therapy for resistance / intolerance to hydroxyurea, according to the prescription criteria approved in Italy. Patients already on treatment (retrospective part) at the start date of the study and patients included after the start date for a period of 9 months may be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
effectiveness of ruxolitinib | at 3 months
  Proportion of patients who reach the target hct <45% within 3 months in the absence of phlebotomy

CONTACTS AND LOCATIONS:
Overall Officials: Paola Guglielmelli, Principal Investigator — AOU Careggi, University of Florence